CLINICAL TRIAL: NCT04389255
Title: Developing a Balance Assessment System With Inertial Sensors and Investigating Validity and Reliability
Brief Title: Developing a Balance Assessment System
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.274
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2019-03

CONDITIONS: Healthy People; Assessment
Keywords: balance; evaluation; İnertial Measurement Unit; validity and reliability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy people: 65 people will be included.
  Interventions: Other: Star Excursion Balance Test; Device: Balance Master device

INTERVENTIONS:
Other: Star Excursion Balance Test — The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals. The test can be used to assess physical performance, but can also be used to screen deficits in dynamic postural control due to musculoskeletal injuries (e.g. chronic ankle instability), to identify athletes at greater risk for lower extremity injury, as well as during the rehabilitation of orthopeadic injuries in healthy active adults.[
Device: Balance Master device — The Balance Master (Neurocom International, Inc Clackamas,) device is a computerized posturography device. The device consists of a fixed support surface consisting of a force table and individuals, a variety of ground elements and a computer screen that will provide visual feedback and conduct test protocols. Posturography tests a person's ability to integrate visual, vestibular and somatosensory inputs and suppress inappropriate sensory information. Thus, it can quantitatively score the person's balance and examine balance problems in detail with the tests it contains. There are various protocols that evaluate balance differently in Balance Master (BMc). Limits of Stability Test (LOS) and Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) were used in the BMc.

SUMMARY:
To develop a balance device that will work with the inertia sensor to quantitatively assess the balance of individuals and investigate the validity and reliability of the balance data of the device.

DETAILED DESCRIPTION:
In this study, we aim to develop a balance assessment system that will measure the balance quantitatively. For this balance assessment system, a balance board will be developed that will work with inertial sensors and detect the oscillations of the individual trying to stand on balance. The validity and reliability of the balance score determined by the analysis of the oscillation data of this balance board will be investigated.

Our hypothesis is that the correlation between the balance score revealed by the newly developed evaluation system and the results of clinical and instrumental balance assessment methods will be significant. For this, one commonly used clinic and one instrumental balance assessment method will be used. Star Excursion Balance Test as a clinical balance assessment method and Balance Master device (BMc) as an instrumental balance assessment method were evaluated. Limits of Stability Test (LOS) and Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) were used in the BMc.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 25
* No neurological or orthopedic diagnosis to affect balance
* Lack of vision and hearing defects that will affect the tests

Exclusion Criteria:

* Existence of refraction problem, visual problem
* Failure to complete the specified tests
* Participant's failure to comply with the study plan

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 65 healthy people, between 18 - 25 years of age
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Newly Developed Balance Assessment System | Day 0
  The newly developed balance evaluation system includes an Arduino based circuit board and an inertial measurement unit consisting of a combination of 3-axis accelerometer and 3-axis gyroscope.
Newly Developed Balance Assessment System | Day 7
  The newly developed balance evaluation system includes an Arduino based circuit board and an inertial measurement unit consisting of a combination of 3-axis accelerometer and 3-axis gyroscope.

SECONDARY OUTCOMES:
Star Excursion Balance Test | Day 0
  The Star Excursion Balance Test (SEBT) is a dynamic test that requires strength, flexibility, and proprioception.
Balance Master device | Day 0
  The Balance Master (Neurocom International, Inc Clackamas,) device is a computerized posturography device.

CONTACTS AND LOCATIONS:
Overall Officials: İlksan Demirbuken, Assoc Prof, Study Chair — Marmara University Health Science Faculty Physiotherapy amd Rehabilitation; Zubeyir Sari, Assoc Prof, Study Director — Marmara University Health Science Faculty Physiotherapy amd Rehabilitation; Ali Omer Acar, Inst, Principal Investigator — Istanbul Aydin University Vocational School of Health Services Physiotherapy
Locations (1):
- Marmara University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cofre Lizama LE, Pijnappels M, Faber GH, Reeves PN, Verschueren SM, van Dieen JH. Age effects on mediolateral balance control. PLoS One. 2014 Oct 28;9(10):e110757. doi: 10.1371/journal.pone.0110757. eCollection 2014. PMID 25350846
- [Background] Corriveau H, Hebert R, Raiche M, Prince F. Evaluation of postural stability in the elderly with stroke. Arch Phys Med Rehabil. 2004 Jul;85(7):1095-101. doi: 10.1016/j.apmr.2003.09.023. PMID 15241756
- [Background] Era P, Sainio P, Koskinen S, Haavisto P, Vaara M, Aromaa A. Postural balance in a random sample of 7,979 subjects aged 30 years and over. Gerontology. 2006;52(4):204-13. doi: 10.1159/000093652. PMID 16849863
- [Background] Suzuki Y, Yatoh S, Suzuki H, Tanabe Y, Shimizu Y, Hada Y, Shimano H. Age-dependent changes in dynamic standing-balance ability evaluated quantitatively using a stabilometer. J Phys Ther Sci. 2018 Jan;30(1):86-91. doi: 10.1589/jpts.30.86. Epub 2018 Jan 27. PMID 29410573
- [Background] Ericksen H, Gribble PA. Sex differences, hormone fluctuations, ankle stability, and dynamic postural control. J Athl Train. 2012 Mar-Apr;47(2):143-8. doi: 10.4085/1062-6050-47.2.143. PMID 22488279
- [Background] Glave AP, Didier JJ, Weatherwax J, Browning SJ, Fiaud V. Testing Postural Stability: Are the Star Excursion Balance Test and Biodex Balance System Limits of Stability Tests Consistent? Gait Posture. 2016 Jan;43:225-7. doi: 10.1016/j.gaitpost.2015.09.028. Epub 2015 Oct 26. PMID 26514832
- [Background] Nakagawa HB, Ferraresi JR, Prata MG, Scheicher ME. Postural balance and functional independence of elderly people according to gender and age: cross-sectional study. Sao Paulo Med J. 2017 May-Jun;135(3):260-265. doi: 10.1590/1516-3180.2016.0325280217. PMID 28746661